CLINICAL TRIAL: NCT05513742
Title: A Phase 2 Study of CTX-009 in Adult Patients With Metastatic Colorectal Cancer Who Have Received Two or Three Prior Systemic Chemotherapy Regimens
Brief Title: A Study of CTX-009 in Adult Patients With Metastatic Colorectal Cancer
Acronym: COMPANION-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Compass Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTX-009-003
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer; Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Approximately 37 patients will be enrolled into Stage 1, and if criteria are met to move to Stage 2, an additional 47 patients will be enrolled, for a total of approximately 84 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX-009 Treatment (Experimental)
  Interventions: Drug: CTX-009

INTERVENTIONS:
Drug: CTX-009 — IV infusion administered on day 1 and 15 of every 28-day cycle

SUMMARY:
This study is designed as an open-label, adaptive Simon Two-Stage study to evaluate the efficacy of CTX-009 in patients with metastatic colorectal cancer.

A Simon Two-Stage adaptive design will enroll approximately 37 patients into Stage 1, and if criteria are met to move to Stage 2, an additional 47 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Histologically or cytologically confirmed metastatic or recurrent colorectal cancers
3. The primary tumor must have been resected > 3 months prior to planned C1D1.
4. Patients who experienced progressive disease or relapse after receiving two or three prior lines of systemic therapy in the locally advanced or metastatic setting. Prior lines of systemic treatment must have included at least one fluoropyrimidine, oxaliplatin, irinotecan, and bevacizumab containing chemotherapy regimen (in any combination and may have been administered in the neoadjuvant setting).

   1. Patients whose tumor is not right sided and RAS wild type must also have received an anti-epidermal growth factor receptor (EGFR) therapy.
   2. Patients with tumors harboring mutations or other alterations for which there are available targeted therapies (e.g. BRAF V600E, HER2-positive, MSI-H/dMMR, etc.) must have also received the relevant approved targeted therapies.
   3. If patient received peri-operative treatment (neoadjuvant and/or adjuvant), please consult the Sponsor Medical Monitor for review of prior treatment lines.
5. At least one lesion measurable as defined by RECIST v1.1
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
7. Predicted life expectancy of at least 12 weeks
8. Adequate hepatic and renal function within 14 days of C1D1 as described below:

   1. Total bilirubin ≤ 1.5 X upper limit of normal (ULN)
   2. Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤ 3.0 X ULN (≤ 5x ULN in case of hepatic metastasis)
   3. Estimated creatinine clearance ≥ 30 mL/min based on Cockcroft-Gault estimated creatinine clearance
   4. Urine protein ≤ 1+ by spot urinalysis (or, if > 1+ then 24 hr urine protein <1.0 g/24 hr)
9. Female patients who are women of childbearing potential (WCBP) must have a negative pregnancy test (serum-human chorionic gonadotropin [hCG] or urine-hCG) at Screening within 14 days of C1D1
10. Female patients must be surgically sterile (or have a monogamous partner who is surgically sterile) or be at least 2 years postmenopausal or commit to use 2 acceptable forms of birth control (defined as the use of an intrauterine device (IUD), a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence) for the duration of the study and for 4 months following the last dose of study treatment. Male patients must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control (condoms with spermicide) for the duration of the study and for 4 months following the last dose of study treatment
11. Signed and dated Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved Informed Consent Form (ICF) before any protocol-directed screening procedures are performed

Exclusion Criteria:

1. From the time point of signed informed consent,

   1. Less than 4 weeks have elapsed since patients had a surgery or major procedure
   2. Less than 2 weeks have elapsed from the last treatment date since patients had any radiation therapy
2. Prior to planned C1D1,

   1. Less than 4 weeks have elapsed since patients had chemotherapy or targeted therapy for colorectal cancer
   2. Less than 4 weeks have elapsed since patients had anticancer immunotherapy or investigational drug treatment
3. A history of the following cardiovascular diseases in past 5 years may be exclusionary, as determined by the Sponsor Medical Monitor:

   1. Congestive heart failure that corresponds to Class II or a higher class under New York Heart Association (NYHA) classification or less than 50% of left ventricular ejection fraction (LVEF)
   2. Uncontrolled hypertension (systolic blood pressure [SBP]/diastolic blood pressure [DBP] > 140/90 mmHg) (e.g., patient with SBP/DBP > 140/90 mmHg despite the best care including anti-hypertensive medications)
   3. Patients with a history of hypertensive crisis or pre-existing hypertensive encephalopathy
   4. Pulmonary hypertension
   5. Myocardial infarction
   6. Uncontrolled arrhythmia
   7. Unstable angina
   8. Patients with any significant vascular diseases (e.g., aortic aneurysm requiring surgery or recent peripheral artery thrombosis) within 6 months prior to the initial treatment of the investigational product
4. Symptomatic or uncontrolled central nervous system (CNS) metastasis (However, patients with asymptomatic CNS metastasis can participate provided that systemic corticosteroid treatment was discontinued at least 4 weeks prior to screening and that the patient is radiologically and neurologically stable or improving)
5. A history of the following hemorrhage-related or gastroenterological disease:

   1. Active hemorrhage, hemorrhagic diathesis, coagulopathy or tumor invasion into great arteries
   2. History of clinically significant and active (within 6 months) gastroenterological disease, such as peptic ulcer, gastrointestinal (GI) bleeding, GI or non-GI fistula, perforation, abdominal abscess, clinical symptoms and signs of GI obstruction, need for parenteral hydration or nutrition, or inflammatory bowel disease.
6. Patients who received antiplatelet drugs (aspirin, clopidogrel, etc.) or anticoagulant drugs (warfarin, heparin, direct thrombin inhibitors, etc.) within 2 weeks prior to C1D1, or are expected to need those drugs during the clinical study.
7. Patients requiring continuous treatment with systemic non-steroidal anti-inflammatory drugs (NSAIDs) or systemic corticosteroids (the following cases are permitted):

   1. NSAIDs: Up to 3 consecutive days' use is permitted
   2. Corticosteroids: Topical use of corticosteroid, such as topical intra-articular injection, intranasal administration, eye drops, inhaler, etc., or temporary systemic corticosteroid use for treatment and prevention of patient's contrast media allergy, or adverse event, is permitted
8. Severe infection requiring systemic antibiotics, antivirus drugs, etc., or other uncontrolled acute active infectious diseases
9. Patients with evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Inactive hepatitis B carriers who tested HBsAg positive may enroll provided that the patient's liver function values are normal. Also, patients with chronic HBV infection which has been controlled by the site's treatment guideline may enroll. HCV patients showing sustained viral response or patients with immunity to HBV infection may enroll
10. Patients with other severe diseases or uncontrolled illnesses that warrant the exclusion from the study (permitted only if medically controlled) including but not limited to:

    1. Pre-existing hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 28 days prior to screening
    2. Major, unhealed injury, active ulcer or untreated fracture
    3. History of cerebrovascular incident (ischemic or hemorrhagic stroke), transient ischemic attack or subarachnoid hemorrhage within 6 months prior to screening
    4. Moderate to severe ascites and/or pleural effusion
11. Clinically significant abnormal electrocardiography (ECG) findings or history determined as clinically significant by the Investigator
12. QT interval (Fridericia's formula) (QTcF) interval > 450 msec at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | From Cycle 1 Day 1 (C1D1) to treatment discontinuation for any reason, average of 6 months
  Percentage of patients whose Best Overall Response (BOR) is assessed as Complete Response (CR) or Partial Response (PR) as assessed by RECIST v1.1

SECONDARY OUTCOMES:
Disease Control Rate | From C1D1 to treatment discontinuation for any reason, average of 6 months
  Percentage of patients whose BOR is assessed as CR, PR, or Stable Disease (SD)
Duration of Response | From first confirmed CR or PR to confirmed PD, average of 6 months
  The time between the date of the radiological evaluation that first confirmed CR or PR and the date of the radiation evaluation that first confirmed Progressive Disease (PD)
Progression Free Survival | From C1D1 to first documented objective PD or death if PD does not occur, average of 6 months
  Time from C1D1 until the date of objective PD (as assessed by RECIST v1.1) or the date of death (by any cause in the absence of disease progression)
Overall Survival | From C1D1 to death from any cause, average of 9 months
  Time from C1D1 until the date of death by any cause. Patients who are still alive at the time of the analysis, or who have become lost to follow-up or withdrawn consent will be censored at their last date known to be alive
Safety Profile of CTX-009 | From C1D1 to 60 days after the last dose of study treatment, average of 7 months
  Incidence of Treatment Emergent Adverse Events (TEAEs) and changes in clinical abnormalities for all randomized patients who received at least one dose of study treatment
Quality of Life Changes | From screening to treatment discontinuation for any reason, average of 6 months
  Assessed approximately every 2 months from patient reported data using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (QLQ)-C30 as compared to baseline responses
Exposure Response by Pharmacokinetic (PK) Sampling | From C1D1 to treatment discontinuation for any reason, average of 6 months
  Serum concentrations of CTX-009 at specified timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Minori Rosales, MD, PhD, Study Director — Compass Therapeutics
Locations (7):
- United States (7):
  - Genesis Cancer and Blood Institute, Hot Springs, Arkansas
  - Florida Cancer Specialists & Research Institute - South, Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute - North, St. Petersburg, Florida
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Zangmeister Cancer Center, Columbus, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided